CLINICAL TRIAL: NCT03474588
Title: Computer Based Training in CBT for Spanish-Speaking Alcohol Users
Brief Title: CBT4CBT With Spanish Alcohol Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000020677; R01AA025605 (NIH)
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (ST) (Active Comparator): This is the same as the treatment normally received at this clinic. This will be tailored to participants' needs, but generally includes individual and group therapy sessions and regular urine monitoring. Sessions will generally last for 1 hour one time per week for 8 weeks and include issues such as:
  * Teaching about the treatment program
  * Teaching important ideas about recovery
  * Increasing knowledge about specific problems about addiction
  * Demonstrating new ways of coping with skills designed to fit each participant
  Interventions: Behavioral: Standard Treatment (ST)
- 2. Standard treatment (ST) PLUS web-based CBT4CBT (Experimental): This is the same as the treatment normally received at this clinic. This will be tailored to participants' needs, but generally includes individual and group therapy sessions and regular urine monitoring. Sessions will generally last for 1 hour one time per week for 8 weeks and include issues such as:
  * Teaching about the treatment program
  * Teaching important ideas about recovery
  * Increasing knowledge about specific problems about addiction
  * Demonstrating new ways of coping with skills designed to fit each participant PLUS
  Participants will have access the CBT4CBT website in Spanish as an add-on to treatment. In this treatment participants will work with a computerized program that teaches skills for stopping alcohol use and increasing coping skills, such as how to understand patterns of alcohol use, how to cope with cravings for alcohol, how to refuse offers of alcohol, and so on.
  Interventions: Behavioral: Standard treatment (ST) PLUS web-based CBT4CBT

INTERVENTIONS:
Behavioral: Standard treatment (ST) PLUS web-based CBT4CBT — Participants will have access to the CBT4CBT website in Spanish as an add-on to treatment. In this treatment participants will work with a computerized program that teaches skills for stopping alcohol use and increasing coping skills, such as how to understand patterns of alcohol use, how to cope with cravings for alcohol, how to refuse offers of alcohol, and so on
  Arms: 2. Standard treatment (ST) PLUS web-based CBT4CBT
Behavioral: Standard Treatment (ST) — ST includes individual and group therapy sessions and regular urine monitoring. Sessions will generally last for 1 hour one time per week for 8 weeks
  Arms: Standard Treatment (ST)

SUMMARY:
Specific aims are as follows:

* To adapt our existing CBT4CBT program for use with Spanish-speaking alcohol users in a web-based platform
* To conduct an 8-week randomized trial evaluating the feasibility and efficacy of adding CBT4CBT-Spanish to treatment as usual in a community based treatment program in a population of 90 Spanish-speaking individuals who meet current criteria for alcohol use disorder
* To evaluate the long-term durability and/or delayed emergence of treatment effects through a six month follow-up after termination of the study treatments. Given previous evidence regarding the durability of standard clinician-delivered CBT and computer-assisted CBT4CBT, we hypothesize that CBT4CBTSpanish will be significantly more effective than standard treatment alone through the follow-up.

DETAILED DESCRIPTION:
The investigators will conduct a Stage 1 randomized clinical trial evaluating the program in which 90 Spanish-speaking individuals with alcohol use disorder will be randomized to (1) standard outpatient counseling at the Hispanic Clinic (ST; typically consisting of weekly individual and group supportive counseling) or (2) CBT4CBT-Spanish as an adjunct to ST. Other aspects of the trial will parallel those in the investogators completed trial of the English version of CBT4CBT-Alcohol to facilitate comparability across studies. Treatments will be delivered over an 8-week period with a 6-month follow-up to assess durability and/or delayed emergence of treatment effects. The primary outcome measure will be percent days of abstinence (PDA) by week. Secondary outcomes include percent heavy drinking days and number of individuals with no heavy drinking days in the last 4 weeks of treatment.

Participants will be 90 individuals seeking treatment for alcohol use at the Hispanic Clinic of CMHC. The clinic treats a heterogeneous population, where 42% of those in the co-occurring treatment program report alcohol as their principal substance related issue and 43% are women. As reported above, the investigators have demonstrated the ability to recruit, randomize, retain, and follow-up high numbers of closely related samples in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 years of age or older.
2. Are applying for outpatient alcohol treatment, with some alcohol use in the past 30 days
3. Speak Spanish as their preferred or principal (most commonly spoken) language.
4. Are sufficiently stable for 8 weeks of outpatient treatment
5. Can commit to 8 weeks of treatment and are willing to be randomized to treatment
6. Are willing to provide locator information for follow-up.

Exclusion Criteria:

1. Have an untreated bipolar or schizophrenic disorder
2. Have a current legal case pending such that incarceration during the 8 week protocol is likely
3. Meet DSM-5 criteria for another current substance use disorder (other than nicotine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Paris, PsyD, Principal Investigator — Yale University
Locations (5):
- United States (5):
  - Midwestern Connecticut Council on Alcoholism (MCCA), Bridgeport, Connecticut
  - Cornell Scott - Hill Health Center, New Haven, Connecticut
  - Hispanic Clinic of CMHC, New Haven, Connecticut
  - Midwestern Connecticut Council on Alcoholism (MCCA), New Haven, Connecticut
  - Multi-Cultural Ambulatory Addiction Services (MAAS), New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benitez B, Frankforter T, Nich C, Paris M, Kiluk BD. Comparing content within a culturally-adapted digital treatment for Hispanic patients with alcohol use disorder. NPJ Digit Med. 2025 Dec 8;9(1):23. doi: 10.1038/s41746-025-02197-7. PMID 41361015

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment (ST): This is the same as the treatment normally received at this clinic. This will be tailored to participants' needs, but generally includes individual and group therapy sessions and regular urine monitoring. Sessions will generally last for 1 hour one time per week for 8 weeks and include issues such as:
  * Teaching about the treatment program
  * Teaching important ideas about recovery
  * Increasing knowledge about specific problems about addiction
  * Demonstrating new ways of coping with skills designed to fit each participant
  Standard Treatment (ST): ST includes individual and group therapy sessions and regular urine monitoring. Sessions will generally last for 1 hour one time per week for 8 weeks
- Standard Treatment (ST) PLUS Web-based CBT4CBT: This is the same as the treatment normally received at this clinic. This will be tailored to participants' needs, but generally includes individual and group therapy sessions and regular urine monitoring. Sessions will generally last for 1 hour one time per week for 8 weeks and include issues such as:
  * Teaching about the treatment program
  * Teaching important ideas about recovery
  * Increasing knowledge about specific problems about addiction
  * Demonstrating new ways of coping with skills designed to fit each participant PLUS
  Participants will have access the CBT4CBT website in Spanish as an add-on to treatment. In this treatment participants will work with a computerized program that teaches skills for stopping alcohol use and increasing coping skills, such as how to understand patterns of alcohol use, how to cope with cravings for alcohol, how to refuse offers of alcohol, and so on.
  Standard treatment (ST) PLUS web-based CBT4CBT: Participants will have access to the CBT4CBT website in Spanish as an add-on to treatment. In this treatment participants will work with a computerized program that teaches skills for stopping alcohol use and increasing coping skills, such as how to understand patterns of alcohol use, how to cope with cravings for alcohol, how to refuse offers of alcohol, and so on
Period: Overall Study
Arm/Group | Standard Treatment (ST) | Standard Treatment (ST) PLUS Web-based CBT4CBT
Started | 28 | 23
Follow up 1 | 27 | 21
Follow up 2 | 27 | 20
Follow up 3 | 25 | 18
Completed | 24 | 19
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment (ST) | Standard Treatment (ST) PLUS Web-based CBT4CBT | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13) | 44.8 (11.9) | 41.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 23 | 51
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 23 | 51
Client Origin of birth [Count of Participants; unit: Participants]
  Client: Puerto Rico | 7 | 7 | 14
  Client: United States | 1 | 1 | 2
  Client: South American country | 1 | 2 | 3
  Client: Mexico | 14 | 6 | 20
  Client: Other Central American country | 5 | 6 | 11
  Client: Carribean Island | 0 | 1 | 1
  Mother: Puerto Rico | 7 | 7 | 14
  Mother: United States | 0 | 0 | 0
  Mother: South American country | 1 | 2 | 3
  Mother: Mexico | 14 | 6 | 20
  Mother: Other Central American country | 6 | 7 | 13
  Mother: Carribean Island | 0 | 1 | 1
  Father: Puerto Rico | 7 | 7 | 14
  Father: United States | 0 | 0 | 0
  Father: South American country | 1 | 2 | 3
  Father: Mexico | 14 | 6 | 20
  Father: Other Central American country | 6 | 7 | 13
  Father: Carribean Island | 0 | 1 | 1
Completed High School [Count of Participants; unit: Participants] | 12 | 12 | 24
Never married/living alone [Count of Participants; unit: Participants] | 15 | 19 | 34
Unemployed [Count of Participants; unit: Participants] | 10 | 9 | 19
On parole or probation [Count of Participants; unit: Participants] | 7 | 8 | 15
Referred by criminal justice system [Count of Participants; unit: Participants] | 7 | 10 | 17
On Public Assistance [Count of Participants; unit: Participants] | 10 | 6 | 16
Previous computer experience [Count of Participants; unit: Participants] | 21 | 12 | 33
Lifetime anxiety disorder [Count of Participants; unit: Participants] | 5 | 6 | 11
Lifetime major depression [Count of Participants; unit: Participants] | 16 | 11 | 27
Lifetime PTSD by SCID [Count of Participants; unit: Participants] | 3 | 7 | 10
Current PTSD by SCID [Count of Participants; unit: Participants] | 3 | 6 | 9
Current anxiety disorder [Count of Participants; unit: Participants] | 4 | 3 | 7
Current major depression [Count of Participants; unit: Participants] | 10 | 11 | 21
Alcohol Use Disorder (AUD) Severity Rating [Count of Participants; unit: Participants] — AUD scale: Mild: The presence of 2 to 3 symptoms, Moderate: The presence of 4 to 5 symptoms, Severe: The presence of 6 or more symptoms.
  Participants
    Mild | 0 | 1 | 1
    Moderate | 7 | 6 | 13
    Severe | 21 | 16 | 37
Diagnosed PTSD by PCL-5 [Count of Participants; unit: Participants] — The PCL-5 is a questionnaire used to assess symptom criteria for PTSD.
  Participants | 5 | 5 | 10
Alcohol Use Disorders Identification Test (Audit) Score 16 or higher [Count of Participants; unit: Participants] — Total score range of 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol. A score of 1 to 7 suggests low-risk consumption, scores from 8 to 14 suggest hazardous or harmful alcohol consumption and a score of 15 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).
  Participants | 18 | 14 | 32
Days paid for work in past 28 [Mean (Standard Deviation); unit: days] | 14.1 (11.6) | 10.7 (10.1) | 12.6 (11)
Days of alcohol use in the past 28 [Mean (Standard Deviation); unit: days] | 9.1 (9.3) | 7.7 (7.3) | 8.5 (8.4)
Days of heavy alcohol use in the past 28 [Mean (Standard Deviation); unit: days] | 7 (8.7) | 5.4 (6.4) | 6.3 (7.7)
Drinks per drinking days in the past 28 [Mean (Standard Deviation); unit: drinks] | 8.6 (5.9) | 10.9 (14.1) | 9.6 (10.4)
Percent days of alcohol abstinence in the past 28 [Mean (Standard Deviation); unit: percentage of days] | 67.5 (33.2) | 72.4 (26.2) | 69.7 (30)
Percent days of heavy drinking in the past 28 [Mean (Standard Deviation); unit: percentage of days] | 25.2 (31.1) | 19.3 (23) | 22.5 (27.6)
Percent days of alcohol abstinence at week 0 [Mean (Standard Deviation); unit: percentage of days] | 73.5 (35.4) | 77 (25.8) | 75.1 (31.1)
Percent days of heavy drinking at week 0 [Mean (Standard Deviation); unit: percentage of days] | 20.4 (32.2) | 14.9 (20.9) | 17.9 (27.5)
Age first used alcohol [Mean (Standard Deviation); unit: years] | 17.1 (4.9) | 17.5 (6.8) | 17.3 (5.8)
Years of alcohol use [Mean (Standard Deviation); unit: years] | 21.1 (13.2) | 25.8 (14.9) | 23.2 (14)
Pre-treatment Alcohol Symptom Count [Mean (Standard Deviation); unit: symptom count] | 7.7 (2.4) | 7.6 (2.6) | 7.7 (2.5)
Pre-treatment AUDIT Score [Mean (Standard Deviation); unit: score on a scale] — Total score range of 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol. A score of 1 to 7 suggests low-risk consumption, scores from 8 to 14 suggest hazardous or harmful alcohol consumption and a score of 15 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).
  score on a scale | 20.3 (9.2) | 18.9 (7.7) | 19.7 (8.5)
Years living in United States [Mean (Standard Deviation); unit: years] | 19.5 (14) | 19.2 (10) | 19.3 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Will be Percent Days of Abstinence (PDA) by Week
Description: The primary outcome measure will be percent days of abstinence (PDA) by week, presented are the raw means at each time point.
Time Frame: By week for 8 weeks
Population: One participant was lost to follow up beginning week 4 in the Standard treatment (ST) PLUS web-based CBT4CBT.
Measure: Mean (Standard Deviation); unit: percentage of days abstinent per week
Arm/Group | Standard Treatment (ST) PLUS Web-based CBT4CBT | Standard Treatment (ST)
Number analyzed (Participants) | 23 | 28
percentage of days abstinent per week
  week 0 (baseline) | 73.29 (25.71) | 66.96 (34.59)
  week 1 | 88.20 (19.57) | 79.59 (30.97)
  week 2 | 83.23 (22.65) | 78.06 (29.22)
  week 3 | 91.30 (11.98) | 77.55 (31.69)
  week 4: number analyzed (Participants) | 22 | 28
  week 4 | 90.26 (15.52) | 71.43 (30.61)
  week 5: number analyzed (Participants) | 22 | 28
  week 5 | 92.86 (12.27) | 72.45 (28.29)
  week 6: number analyzed (Participants) | 22 | 28
  week 6 | 89.61 (14.74) | 80.10 (29.70)
  week 7: number analyzed (Participants) | 22 | 28
  week 7 | 87.01 (24.11) | 77.04 (31.67)
  week 8: number analyzed (Participants) | 22 | 28
  week 8 | 84.42 (22.44) | 75.51 (31.55)
Statistical Analysis 1: Comparison: Standard Treatment (ST) PLUS Web-based CBT4CBT vs Standard Treatment (ST); Test type: Superiority; p = 0.30, Regression, Linear — Presented is the p value for the interaction between time and treatment; Random Effects Regression Models (RERM), time was log transformed to account for expectation of greater change closer to baseline

2. Primary Outcome: Monthly Abstinence From Alcohol
Description: Estimated means of sustained abstinence calculated as percent days per month from month 3 through 8 in post intervention follow up.
Time Frame: Months 3 through 8 (6 months total)
Population: All participants assessed during the period.
Measure: Mean (Standard Deviation); unit: percentage of days abstinent in a month
Arm/Group | Standard Treatment (ST) PLUS Web-based CBT4CBT | Standard Treatment (ST)
Number analyzed (Participants) | 21 | 27
percentage of days abstinent in a month
  month 3 | 89.03 (10.55) | 77.46 (29.30)
  month 4 | 89.85 (10.55) | 76.88 (29.30)
  month 5 | 90.67 (10.55) | 76.31 (29.30)
  month 6 | 91.49 (10.55) | 75.74 (29.30)
  month 7 | 92.30 (10.55) | 75.17 (29.30)
  month 8 | 93.12 (10.55) | 74.59 (29.30)
Statistical Analysis 1: Comparison: Standard Treatment (ST) PLUS Web-based CBT4CBT vs Standard Treatment (ST); Random Effects Regression Model (RERM), included in the model were treatment, time and the interaction of time and treatment; Test type: Superiority; p = 0.14, Regression, Linear — presented is the p value for the interaction of treatment and time in the model; Mean Difference (Net) = 1.39, 95% CI 2-sided [-0.46 to 3.24], Standard Error of Mean 0.94

3. Secondary Outcome: Secondary Outcomes Include Percent Heavy Drinking Days
Description: Percent heavy drinking days during 8 weeks of trial
Time Frame: 8 weeks
Population: Participants completing the full study.
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Standard Treatment (ST) PLUS Web-based CBT4CBT | Standard Treatment (ST)
Number analyzed (Participants) | 22 | 28
percentage of heavy drinking days | 6.4 (10.3) | 15.2 (22.7)
Statistical Analysis 1: Comparison: Standard Treatment (ST) PLUS Web-based CBT4CBT vs Standard Treatment (ST); Test type: Superiority; p = 0.097, ANOVA

4. Secondary Outcome: Number of Individuals With no Heavy Drinking Days in the Last 4 Weeks of Treatment
Description: Number of individuals with no heavy drinking days in the last 4 weeks of treatment
Time Frame: last 4 weeks of treatment (4 weeks)
Population: Participants completing the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment (ST) PLUS Web-based CBT4CBT | Standard Treatment (ST)
Number analyzed (Participants) | 22 | 28
Participants | 11 | 13
Statistical Analysis 1: Comparison: Standard Treatment (ST) PLUS Web-based CBT4CBT vs Standard Treatment (ST); Test type: Superiority; p = 0.802, Chi-squared

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Standard Treatment (ST) | Standard Treatment (ST) PLUS Web-based CBT4CBT
All-Cause Mortality (participants affected / at risk) | 0/28 | 1/23
Serious Adverse Events (participants affected / at risk) | 2/28 | 4/23
Other Adverse Events (participants affected / at risk) | 0/28 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment (ST) (N=28) | Standard Treatment (ST) PLUS Web-based CBT4CBT (N=23)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (2) | 0 (0) — Hospitalization for Alcohol Use symptoms
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Hospitalization for Detox
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) — Hospitalization for Mental health
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 2 (2) — Hospitalization for Infection
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1) — Hospitalization for Kidney stones

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03474588/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03474588/SAP_002.pdf
  • Informed Consent Form (2021-09-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT03474588/ICF_000.pdf